CLINICAL TRIAL: NCT00947323
Title: The Effect of Simvastatin in the Penile Erection: a Randomized, Double-blind Clinical Trial
Brief Title: Simvastatin for Treating Erectile Dysfunction
Acronym: STED
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Santa Casa de Porto Alegre (Other)
Responsible Party: Eduardo Touguinha Mastalir, Santa Casa de Porto Alegre
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: STED
Record Dates: First submitted 2009-07-27; First posted 2009-07-28 (Estimated); Last update posted 2010-09-27 (Estimated); Status verified 2010-09

CONDITIONS: Erectile Dysfunction; Vascular Disease Detected; C Reactive Protein
Keywords: simvastatin; endothelial dysfunction; erectile dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Simvastatin (Experimental): Treatment arm.
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Simvastatin — simvastatin 20 daily for six months.
  Arms: Simvastatin
Drug: Placebo
  Arms: placebo

SUMMARY:
This is a randomized clinical trial, double-blind, placebo controlled, to verify if simvastatin can improve erectile dysfunction in men with endothelial dysfunction, without any cardiac disease.It is hypothesized that the simvastatin can improve the endothelial function, improving the nitric oxide liberation in corpora cavernosa of the penis, resulting in improvement of erection.

ELIGIBILITY:
Inclusion Criteria:

* Erectile dysfunction
* Elevated C reactive protein
* Able to adhere the protocol

Exclusion Criteria:

* Diabetes mellitus
* Cardiac disease
* Cerebral vascular disease
* Hypogonadism
* Any contraindication to simvastatin

Ages: 35 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2006-01; Primary Completion 2008-07 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Penile erection